CLINICAL TRIAL: NCT04208399
Title: A Single-Dose, Open-Label, Parallel-Group Study to Evaluate the Effect of Hepatic Impairment on the Pharmacokinetics of JNJ-56136379
Brief Title: A Study to Evaluate the Effect of Hepatic Impairment on JNJ-56136379
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Sciences Ireland UC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR108713; 2019-003071-20 (EudraCT Number); 56136379HPB1009 (Other: Janssen Sciences Ireland UC)
Record Dates: First submitted 2019-12-20; First posted 2019-12-23 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Hepatic Impairment
MeSH Terms: interventions — JNJ-56136379

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Part A: Group 1 (Experimental): Participants with liver cirrhosis with moderate hepatic impairment will receive a single oral dose of JNJ-56136379 in fed condition.
  Interventions: Drug: JNJ-56136379
- Part A: Group 2 (Experimental): Participants with normal liver function with no liver cirrhosis will receive a single oral dose of JNJ-56136379 in fed condition.
  Interventions: Drug: JNJ-56136379
- Part B: Group 3 (optional) (Experimental): Participants with liver cirrhosis with mild hepatic impairment will receive a single oral dose of JNJ-56136379 in fed condition.
  Interventions: Drug: JNJ-56136379
- Part B: Group 4 (optional) (Experimental): Participants with liver cirrhosis with severe hepatic impairment will receive a single oral dose of JNJ-56136379 in fed condition.
  Interventions: Drug: JNJ-56136379

INTERVENTIONS:
Drug: JNJ-56136379 — JNJ-56136379 will be administered orally in fed condition.

SUMMARY:
The purpose of the study is to evaluate the pharmacokinetics (PK) of a single oral dose of JNJ-56136379 in participants with liver cirrhosis and impaired hepatic function when compared with healthy participants with normal hepatic function and no liver cirrhosis.

ELIGIBILITY:
Inclusion criteria:

* For all participants: Body mass index (BMI) between 18.0 and 38 kilogram per meter square (kg/m2), extremes included; Woman of childbearing potential must not be pregnant; Highly effective contraceptive measures in place for female participants of childbearing potential or male participants with female partners of childbearing potential; Non-smoker or light smoker as defined per protocol.
* For Healthy Participants with Normal Hepatic Function and No Liver Cirrhosis: Demographically comparable to the study groups with hepatic impairment with respect to sex, age (+/-10 years), and body weight (+/-10 kilogram [kg]); Participants must be in good health clinically and biologically as defined per protocol.
* For Participants with Liver Cirrhosis and Moderate or Mild or Severe Hepatic Impairment: Must have a total Child-Pugh score of 5 or 6, inclusive (mild); or 7 to 9, inclusive (moderate); or 10 to 15, inclusive (severe) as determined by the investigator; Must have liver cirrhosis with fibro scan readout greater than (>) 12.5 Kilopascal (kPa) as cut-off at screening
* Participants with controlled hypertension, with problems directly associated with the primary diagnosis of hepatic impairment and with concurrent stable medical conditions if the condition(s) will not introduce an additional risk factor and will not interfere with the study objectives.
* Concomitant medications to treat underlying disease states or medical conditions related to hepatic impairment are allowed.

Exclusion Criteria:

* History of / or current clinically significant medical illness that could interfere with the interpretation of the study results.
* Known allergies, hypersensitivity, or intolerance to JNJ-6379 or its excipients.
* History of drug or alcohol abuse within 1 year before screening or positive test results at screening and Day -1.
* Blood or blood products donated or substantial loss of blood (more than 500 milliliters [mL]) within 3 months before the study starts
* Experimental drug received (including investigational vaccines) or experimental medical device used within 1 month or within a period less than 10 times the drug's half-life, whichever is longer, before the first dose of the study intervention is scheduled.
* Evidence of infection with human immunodeficiency virus (HIV)-1 and HIV-2, hepatitis A, B or C (except if sustained virologic response to hepatitis C virus [HCV] treatment).
* Inability to fast for 10 hours.
* Signs of hepatocellular carcinoma or history of biliary obstruction within the past 2 years.
* Lack of good or reasonable venous access.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-01-09 (Actual); Primary Completion 2021-03-26 (Actual); Study Completion 2021-03-26 (Actual)

PRIMARY OUTCOMES:
Plasma Concentration of JNJ-56136379 | Up to Day 21
  Plasma concentration of oral dose of JNJ-56136379 will be assessed.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Up to 6 months
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Sciences Ireland UC Clinical Trials, Study Director — Janssen Sciences Ireland UC
Locations (1):
- APEX GmbH, München, Germany

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency